CLINICAL TRIAL: NCT01359748
Title: Clinical Study About Blood Pressure Measurement Efficacy on Multifunction KEITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aguiflai Iberica, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: K8-BP-31032011
Record Dates: First submitted 2011-05-16; First posted 2011-05-25 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Blood Pressure
Keywords: Non Invasive Blood Pressure measurement study.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Wrist Size <= 14.25 Cm (Other): * Blood pressure measured using the reference sphygmomanometer.
  * Blood pressure measured using the Sphygmomanometer under test.
  Interventions: Device: Reference sphygmomanometer; Device: Sphygmomanometer under test
- Wrist Size >=14.26 <16.50 Cm (Other): * Blood pressure measured using the reference sphygmomanometer.
  * Blood pressure measured using the Sphygmomanometer under test.
  Interventions: Device: Reference sphygmomanometer; Device: Sphygmomanometer under test
- Wrist size >=16.5 <17.75 Cm (Other): * Blood pressure measured using the reference sphygmomanometer.
  * Blood pressure measured using the Sphygmomanometer under test.
  Interventions: Device: Reference sphygmomanometer; Device: Sphygmomanometer under test
- Wrist Size >=17.75 Cm (Other): * Blood pressure measured using the reference sphygmomanometer.
  * Blood pressure measured using the Sphygmomanometer under test.
  Interventions: Device: Reference sphygmomanometer; Device: Sphygmomanometer under test

INTERVENTIONS:
Device: Reference sphygmomanometer — * USED Audible Korotkoff (K5)for Auscultatory sphygmomanometer.
  Other Names: *Ref Auscult. sphygm.: RIESTER MINIMUS S/N 20534567
Device: Sphygmomanometer under test — Electronic Oscillometric method.
  Other Names: * Multifunction KEITO K7 S/N 1941.

SUMMARY:
The purpose of this trial is to determine the accuracy of the Blood Pressure (BP) measurement of multifunction KEITO devices under test requirements of the Standard American National Standards Institute(ANSI)/Association for the Advancement of Medical Instrumentation(AAMI)/International Organization for Standardization (ISO): ANSI/AAMI/ISO 81060-2:2009.

DETAILED DESCRIPTION:
Nowadays is important controlling our basic health parameters. Due this, the multifunction KEITO Devices was designed to offer to the general public a convenient way to do so easily in the public sites.

One of the most important parameter is the Blood Pressure (BP)measurement. To warrant their efficacity and accuracy, was essential to perform this trial to ensure that the measurements obtained meet with the requirements of the specific U.S. standard about Non-invasive sphygmomanometers.

By Validating with auscultatory reference sphygmomanometer, as defined on the ANSI/AAMI/ISO 81060-2:2009 , we have been intending to demonstrate that the multifunction KEITO devices, particularly about the Blood Pressure (BP) Measurement, have the same efficacy and accuracy as the conventional auscultatory sphygmomanometers.

To include most of the groups of Blood Pressure (BP) measurements types on this clinical trial, a great variety of BP ranges have been selected, always in accordance with the standard.

ELIGIBILITY:
Inclusion Criteria:

* Wrist circumference: 12 to 20 Cm
* At least 5% of the readings shall have Systolic BP<=100 mmHg
* At least 5% of the readings shall have Systolic BP>=160 mmHg
* At least 20% of the readings shall have Systolic BP>=140 mmHg
* At least 5% of the readings shall have Diastolic BP<=60 mmHg
* At least 5% of the readings shall have Diastolic BP>=100 mmHg
* At least 20% of the readings shall have Diastolic BP>=85 mmHg

Exclusion Criteria:

* Pregnant Women

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel P Ferre, Engineer, Study Director; Francisco B Contreras, Technician, Study Chair

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To recruit the volunteers, we have complied with the limb size distribution required on Standard Association for the American National Standards Institute(ANSI)/Association for the Advancement of Medical Instrumentation (AAMI)/International Organization for Standardization (ISO): ANSI/AAMI/ISO 81060-2:2009 [5.1.4]
Groups:
- Subjects With Wrist Size >=14.26Cm; Subjects With Wrist Size <=14.25Cm; Subjects With Wrist Size >=16.50Cm; Subjects With Wrist Size >=17.75Cm: Patients who meet with chapter 5 of Standard ANSI/AAMI/ISO 81060-2:2009. The reference Aneroid sphygmomanometer RIESTER MINIMUS II has an adjustable cuff from 24 cm to 32 cm on arm circumference.
  The KEITO's cuff is not adjustable, the wrist circumference admissible is 12 to 20 cm.
Period: Overall Study
Arm/Group | Subjects With Wrist Size >=14.26Cm | Subjects With Wrist Size <=14.25Cm | Subjects With Wrist Size >=16.50Cm | Subjects With Wrist Size >=17.75Cm
Started | 48 | 20 | 10 | 11
Completed | 48 | 20 | 10 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Wrist Size <=14.25Cm; Wrist Size<=16.40 Cm; Wrist Size >=16.5 Cm; Wrist Size >=17.75: Subjects, males or females, with wrist size specified.
- Total: Total of all reporting groups
Arm/Group | Wrist Size <=14.25Cm | Wrist Size<=16.40 Cm | Wrist Size >=16.5 Cm | Wrist Size >=17.75 | Total
Number analyzed (Participants) | 20 | 48 | 10 | 11 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 14 | 43 | 9 | 10 | 76
  >=65 years | 5 | 5 | 1 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 26 | 1 | 2 | 41
  Male | 8 | 22 | 9 | 9 | 48

OUTCOME MEASURES:

1. Primary Outcome: BP Measurements Using the Reference Auscultatory Sphygmomanometer
Description: The subject was measured by the two observers at the same time using the reference sphygmomanometer and double stethoscope.
  The observers agree to take the K5 korotkoff sound. Each observer takes notes of their own measures.
Time Frame: Five minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Subjects: Subjects who meet with chapter 5 of Standard ANSI/AAMI/ISO 81060-2:2009
Arm/Group | Subjects
Number analyzed (Participants) | 89
mmHg
  Systolic Maximum (mmHg) | 186 (3.1)
  Diastolic Maximum (mmHg) | 107 (3.0)
  Systolic Minimum (mmHg) | 93 (3.1)
  Diastolic Minimum (mmHg) | 53 (3.0)

2. Primary Outcome: BP Measurement Using Multifunction KEITO
Description: Prior starting the measurement phase using Multifunction KEITO, the under test device was reset before each new measurement.
  The subject has to be at rest at least 60 seconds before be measured.
Time Frame: 30 seconds
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Subjects: Patients who meet with chapter 5 of Standard ANSI/AAMI/ISO 81060-2:2009
Arm/Group | Subjects
Number analyzed (Participants) | 89
mmHg
  Systolic Maximum | 174 (5.2)
  Diastolic Maximum | 98 (4.5)
  Systolic Minimum | 94 (5.2)
  Diastolic Minimum | 55 (4.5)

ADVERSE EVENTS:
Time Frame: No adverse events were collected.
Description: No adverse events were collected.
Groups:
- Wrist Size <=14.25 Cm: Subjects with wrist size equal or less than 14.25 Cm
- Wrist Size <=16.4Cm: Subjects with wrist size equal or less than 16.40 Cm
- Wrist Size >=16.5 Cm: Subjects with wrist size equal or higher than 16.5 Cm
- Wrist Size >=17.75 Cm: Subjects with wrist size equal or higher than 17.75 Cm
Arm/Group | Wrist Size <=14.25 Cm | Wrist Size <=16.4Cm | Wrist Size >=16.5 Cm | Wrist Size >=17.75 Cm
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/48 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/20 | 0/48 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No